CLINICAL TRIAL: NCT03050814
Title: A Randomized Phase II Trial of Standard of Care Alone or in Combination With Ad-CEA Vaccine and Avelumab in Patients With Previously Untreated Metastatic or Unresectable Colorectal Cancer
Brief Title: Standard of Care Alone or in Combination With Ad-CEA Vaccine and Avelumab in People With Previously Untreated Metastatic Colorectal Cancer QUILT-2.004
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated after an unplanned interim efficacy analysis.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julius Strauss, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170057; 17-C-0057
Record Dates: First submitted 2017-02-10; First posted 2017-02-13 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Tumors; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Adenocarcinoma; Colorectal Cancer
Keywords: Anti-PDL1 Antibody; Therapeutic Cancer Vaccine; Mismatch Repair Deficiency; Progression Free Survival; Adenovirus Based, CEA-Targeting Vaccine
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — avelumab; Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) - Arm A (Active Comparator): Participants will receive leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX)- + bevacizumab + for up to 12 2-week cycles followed by maintenance therapy with bevacizumab + capecitabine until disease progression.
  Interventions: Drug: Bevacizumab; Drug: 5-Fluorouracil (FU); Drug: Leucovorin; Drug: Oxaliplatin; Drug: Capecitabine
- Standard of Care (SOC) - Arm B + Lead in (Experimental): Participants will receive leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX)- + bevacizumab + avelumab + Ad-CEA vaccine (given weeks 0,2,4,8,12,16 and then every 12 weeks) for up to 12 2-week cycles followed by maintenance therapy with bevacizumab + capecitabine + avelumab + Ad-CEA vaccine (following the every 12-week dosing schedule) until disease progression.
  Interventions: Drug: Avelumab; Biological: Ad-CEA vaccine; Drug: Bevacizumab; Drug: 5-Fluorouracil (FU); Drug: Leucovorin; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Avelumab — 10 mg/kg intravenous (IV) over 30-60 min on Day 1
  Other Names: Bavencio
  Arms: Standard of Care (SOC) - Arm B + Lead in
Biological: Ad-CEA vaccine — Subcutaneous injection in the thigh prior to Avelumab on Day 1 of cycles 1, 2 3, 5, 7, 9; every 6 cycles thereafter.
  Arms: Standard of Care (SOC) - Arm B + Lead in
Drug: Bevacizumab — 5mg/kg intravenous (IV) over 30-90 min on day 1 (Arm A) or 2 (Arm B). Part of the standard of care therapy.
  Other Names: Avastin
Drug: 5-Fluorouracil (FU) — 400mg/m^2 (only Arm A) intravenous (IV) bolus on day 1. Part of the standard of care therapy.
  Other Names: Tolak
Drug: Leucovorin — 400mg/m^2 intravenous (IV) over 2 hours on day 1 (Arm A) or Day 2 (Arm B). Part of the standard of care therapy.
  Other Names: folinic acid
Drug: Oxaliplatin — 85mg/m^2 (Arm A) or 68mg/m^2 (Arm B) intravenous (IV) over 2 hours on day 1 (Arm A) or Day 2 (Arm B). Part of the standard of care therapy.
  Other Names: Eloxatin
Drug: Capecitabine — 625 mg/m^2 twice a day by mouth. Part of the standard of care therapy.
  Other Names: Xeloda
Drug: 5-Fluorouracil (FU) — 2400 mg/m^2 (Arm A and B) intravenous (IV) over 46 hours (+/-2 hours) to start on Day 1 (ARM A) or Day 2 (Arm B). Part of the standard of care therapy.
  Other Names: Tolak

SUMMARY:
Background:

Colorectal cancer is a common cancer in the Unites States (U.S.) It causes the second most cancer-related deaths. The drug avelumab and vaccine Ad-CEA together help the immune system fight cancer.

Objective:

To test if avelumab and Ad-CEA plus standard therapy treats colorectal cancer that has spread to other sites better than standard therapy alone.

Eligibility:

People ages 18 and older with untreated colorectal cancer that has spread in the body

Design:

Participants will be screened with:

Test to see if their cancer has a certain deficiency

Blood, urine, and heart tests

Scans

Medical history

Physical exam

Tumor sample. This can be from a previous procedure.

A small group of participants will get Ad-CEA and avelumab plus standard therapy. This is leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX) plus bevacizumab for up to 24 weeks then capecitabine plus bevacizumab.

The others will have treatment in 2-week cycles. They will be Arm A or B:

Arm A: FOLFOX and bevacizumab by intravenous (IV) days 1 and 2 for 12 cycles. After that, capecitabine by mouth twice a day and bevacizumab by IV on day 1.

Arm B: Ad-CEA injection every 2-12 weeks. Avelumab by IV on day 1 of each cycle. FOLFOX and bevacizumab by IV days 2 and 3 for 12 cycles. Then, capecitabine by mouth twice a day and bevacizumab through IV on day 2.

Participants will repeat screening tests during the study.

Participants will be treated until their disease gets worse or they have bad side effects. Arm A participants can join Arm B. They will have a visit 4 5 weeks after they stop therapy.

DETAILED DESCRIPTION:
Background

* Colorectal cancer (CRC) is the fourth most common cancer diagnosis in the United States and accounts for the second most cancer-related deaths.
* Programmed death ligand 1 (PD-L1) is a transmembrane protein that was first identified for its role in the maintenance of self-tolerance and prevention of autoimmunity. Blockade of the interaction between PD-L1 on tumor cells and PD-1 on T cells is expected to reverse T cell suppression within tumors. These agents are dependent on underlying T cell activation against the tumor cell to be effective.
* Avelumab is a fully human immunoglobulin G 1 (IgG1) anti-PDL1 antibody that selectively binds to PD-L1 and competitively blocks its interaction with PD-1.
* In ongoing phase 1 trials of avelumab, the agent has been well tolerated and has shown clinical activity.
* Clinical trials with anti-PD-1/L1 agents in colorectal cancer have resulted in minimal activity in patients who do not have mismatch repair deficiency (MMR-D).
* Therapeutic cancer vaccines targeting overexpressed proteins offer a potential method to activate T cells against tumors.
* A novel adenovirus-based, carcinoembryonic antigen (CEA)-targeting vaccine has demonstrated cytolytic T cell responses in patients with metastatic colorectal cancer.
* Standard of care agents in first line metastatic colorectal cancer (CRC) have properties been associated with improved immune response via immunologic cell death and immunogenic modulation.

Primary Objective

-To determine if there is an improvement progression free survival among patients with metastatic colorectal cancer lacking a mismatch repair deficiency who are treated with standard of care + anti- PDL1 monoclonal antibody + Ad-CEA therapeutic cancer vaccine compared with standard of care alone.

Eligibility

* Subject's age 18 and older with previously untreated pathologically confirmed metastatic or unresectable colorectal cancer; prior adjuvant therapy is acceptable.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Normal organ and bone marrow function.
* Subjects with active autoimmune diseases requiring treatment and subjects requiring system steroids (except for physiologic doses for steroid replacement) are not allowed.
* Tumor sample and whole blood sample must be available for proteomics, genomics and transcriptomics analyses.
* Subjects with metastatic or unresectable colorectal cancer with mismatch repair deficiency (MMR-D or microsatellite instability (MSI)-High) will not be eligible.

Design

* This is a randomized, multicenter phase II clinical trial designed to evaluate the potential improvement in progression free survival (PFS) when Avelumab and Ad-CEA vaccine are used in combination with standard of care therapy in metastatic or unresectable colorectal cancer when compared with standard of care alone (FOLFOX-A).
* A lead in cohort, comprising the first 6 evaluable subjects enrolled, will be treated with avelumab + Ad- CEA vaccine + standard of care in order to assess the safety of the combination.
* If no more than 1 subject in the lead in cohort experiences a dose limiting toxicity attributable to the investigational new drug (IND) agents, 70 evaluable subjects will be randomized on a 1:1 basis to receive either Avelumab + Ad-CEA vaccine + standard of care (Arm B) or standard of care alone (Arm A).
* Standard of care therapy consists of 6 - 12 two-week cycles of bevacizumab + FOLFOX (5-FU, leucovorin, oxaliplatin) followed by two-week cycles of bevacizumab + capecitabine until disease progression.
* Subjects assigned to Arm A that have progressive disease will be offered Avelumab + Ad-CEA vaccine in combination with a standard chemotherapy regimen.
* Kaplan-Meier curves and a two-tailed log-rank test will be the primary analysis methods.
* The accrual ceiling for the study is set at 97.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must have previously untreated metastatic or unresectable colorectal cancer and have no contraindications to treatment with the standard of care regimen as determined by the investigator. Prior adjuvant therapy for surgically resectable disease (including oligometastatic disease) is acceptable (including immunotherapy) but must have been completed at least 6 months prior to enrollment.
* Patients should not be eligible for potentially curative surgical intervention in the case of oligometastatic disease at the time of enrollment or must have actively refused after explicit discussion of potential benefit of this intervention with multidisciplinary team.
* Histologically confirmed colorectal cancer
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Age greater than or equal to 18 years. Because safety data is not known with this agent in patients less than 18 years old, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Patients must have normal organ and marrow function as defined below:

  * Creatinine clearance (per Institutional standard or 24-hour urine) greater than or equal to 30 mL/min.
  * Adequate hepatic function defined by a total bilirubin level less than or equal to 1.5 the upper limit of normal range (ULN), an aspartate aminotransferase (AST), level less than or equal to 2.5 ULN, and an alanine aminotransferase (ALT) level less than or equal to 2.5 ULN or, for subjects with documented metastatic disease to the liver, AST and ALT levels less than or equal to 5 ULN.
  * Hematological eligibility parameters (within16 days of enrollment):
  * Granulocyte count greater than or equal to 1,500/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Hemoglobin greater than or equal to 9 g/dL
* The effects of Ad-CEA vaccine and Avelumab on the developing human fetus are unknown. For this reason and because Ad-CEA vaccine and Avelumab as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for a period of 4 months after the last treatment with avelumab or 6 months after the last administration of bevacizumab, whichever occurs later. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Metastatic or unresectable colorectal cancer with mismatch repair deficiency (MMR-D or microsatellite instability (MSI)-High).
* Concurrent treatment for cancer except agents specified within the treatment protocol.
* Prior surgery or gastrointestinal perforation within 28 days of enrollment.
* Persisting toxicity related to prior therapy (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Grade > 1); however, alopecia, sensory neuropathy Grade <=2, or other Grade <=2 AEs not constituting a safety risk based on investigator's judgment are acceptable.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses less than or equal to 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication).
* Patients who are receiving any other investigational agents within 28 days before start of study treatment.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Subjects with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy. Subjects with CNS metastases incidentally detected during Screening which do not cause clinical symptoms and for which standard of care suggests no therapeutic intervention is needed are eligible.
* Active infection, requiring systemic therapy,
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 3 months prior to enrollment), myocardial infarction (< 3 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or uncontrolled arrhythmias.
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Pregnant women and breastfeeding mothers are excluded due to unknown impact on embryos or infants.
* Known alcohol or drug abuse.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade greater than or equal to 3).
* Patients with a known hypersensitivity/allergy to any of the standard of care agents used in this study or related compounds (e.g., platinum compounds) are excluded.
* Prior history of hypertensive emergency or hypertensive encephalopathy (for those expected to receive bevacizumab.
* Serious, non-healing wound, active ulcer, or untreated bone fracture, including tumor related pathological fracture.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Patients being treated with medications with drug-drug interactions with study agents will require evaluation by to determine if full doses of all study treatments can be given safely. Significant drug-drug interactions will need to be addressed prior to enrollment. Alternatively, the patient will not be eligible.
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Y Strauss, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morse MA, Chaudhry A, Gabitzsch ES, Hobeika AC, Osada T, Clay TM, Amalfitano A, Burnett BK, Devi GR, Hsu DS, Xu Y, Balcaitis S, Dua R, Nguyen S, Balint JP Jr, Jones FR, Lyerly HK. Novel adenoviral vector induces T-cell responses despite anti-adenoviral neutralizing antibodies in colorectal cancer patients. Cancer Immunol Immunother. 2013 Aug;62(8):1293-301. doi: 10.1007/s00262-013-1400-3. Epub 2013 Apr 30. PMID 23624851
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Balint JP, Gabitzsch ES, Rice A, Latchman Y, Xu Y, Messerschmidt GL, Chaudhry A, Morse MA, Jones FR. Extended evaluation of a phase 1/2 trial on dosing, safety, immunogenicity, and overall survival after immunizations with an advanced-generation Ad5 [E1-, E2b-]-CEA(6D) vaccine in late-stage colorectal cancer. Cancer Immunol Immunother. 2015 Aug;64(8):977-87. doi: 10.1007/s00262-015-1706-4. Epub 2015 May 9. PMID 25956394
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0057.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC) - Arm A: Participants will receive leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX)- + bevacizumab + for up to 12 2-week cycles followed by maintenance therapy with bevacizumab + capecitabine until disease progression.
  Bevacizumab: 5mg/kg intravenous (IV) over 30-90 min on day.
  5-Fluorouracil (FU): 400mg/m^2 intravenous (IV) bolus on day 1.
  Leucovorin: 400mg/m^2 intravenous (IV) over 2 hours on day 1.
  Oxaliplatin: 85mg/m^2 intravenous (IV) over 2 hours on day 1.
  Capecitabine: 625 mg/m^2 twice a day by mouth. 5-Fluorouracil (FU): 2400 mg/m^2 intravenous (IV) over 46 hours (+/-2 hours) to start on Day 1.
- Standard of Care (SOC) - Arm B + Lead in: Participants will receive leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX)- + bevacizumab + avelumab + Ad-CEA vaccine (given weeks 0,2,4,8,12,16 and then every 12 weeks) for up to 12 2-week cycles followed by maintenance therapy with bevacizumab + capecitabine + avelumab + Ad-CEA vaccine (following the every 12-week dosing schedule) until disease progression.
  Avelumab: 10 mg/kg intravenous (IV) over 30-60 min on day 1
  Ad-CEA vaccine: Subcutaneous injection in the thigh prior to Avelumab on Day 1 of cycles 1, 2 3, 5, 7, 9; every 6 cycles thereafter.
  Bevacizumab: 5mg/kg intravenous (IV) over 30-90 min on day 2.
  Leucovorin: 400mg/m^2 intravenous (IV) over 2 hours on day 2.
  Oxaliplatin: 68mg/m^2 intravenous (IV) over 2 hours on day 2.
  Capecitabine: 625 mg/m^2 twice a day by mouth.
  5-Fluorouracil (FU): 2400 mg/m^2 intravenous (IV) over 46 hours (+/-2 hours) to start on day 2.
- Enrolled But Not Assigned to a Treatment Arm: 4 participants were enrolled but not treated on Arm A or Arm B. Only baseline data were captured.
Period: Overall Study
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in | Enrolled But Not Assigned to a Treatment Arm
Started | 10 | 16 | 4
Completed | 10 | 16 | 0
Not Completed | 0 | 0 | 4
Not completed — Screen failures | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: 4 participants that were enrolled but not assigned to a treatment arm had baseline data collected and it is reported in this table. These participants were screen failures who were not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in | Enrolled But Not Assigned to a Treatment Arm | Total
Number analyzed (Participants) | 10 | 16 | 4 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.94 (10.65) | 56.34 (8.45) | 59.17 (23.3) | 57.82 (14.13)
Age, Customized [Count of Participants; unit: Participants]
  <= 18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 2 | 23
  >= 65 years | 1 | 4 | 1 | 6
  Missing | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 3 | 15
  Male | 3 | 11 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 15 | 4 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 7
  White | 6 | 13 | 3 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 16 | 4 | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Between the Standard of Care (SOC) Arm A, and Standard of Care (SOC) Arm B + lead-in
Description: Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Up to 1.5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in
Number analyzed (Participants) | 10 | 16
Months | 8.8 [3.3 to 17.0] | 10.1 [3.6 to 16.1]
Statistical Analysis 1: Comparison: Standard of Care (SOC) - Arm A vs Standard of Care (SOC) - Arm B + Lead in; Test type: Other; p = 0.91, Kaplan Meier; Kaplan-Meier curves and a two-tailed log-rank test; Hazard Ratio (HR) = 1.061, 95% CI 2-sided [0.380 to 2.966]

2. Secondary Outcome: Number of Participants That Are Hospitalized Because of Adverse Events Attributed to Disease Progression
Description: Participants hospitalized because of adverse events measured by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 attributed to disease progression. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Up to 51.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in
Number analyzed (Participants) | 10 | 16
Participants | 4 | 4

3. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 33 months and 20 days for Arm A and 51 months and 7 days for Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in
Number analyzed (Participants) | 10 | 16
Participants | 10 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 33 months and 20 days for Arm A and 51 months and 7 days for Arm B.
Arm/Group | Standard of Care (SOC) - Arm A | Standard of Care (SOC) - Arm B + Lead in
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/16
Serious Adverse Events (participants affected / at risk) | 9/10 | 10/16
Other Adverse Events (participants affected / at risk) | 10/10 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) - Arm A (N=10) | Standard of Care (SOC) - Arm B + Lead in (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, coronary vasospasm (Cardiac disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, ureter (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, anuric renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Cystoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (2) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) — Exploratory Lap, converted to partial proctectomy
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) — Exploratory Lap, sigmoidectomy and colostomy
Surgical and medical procedures - Other, Hepatic RFA, Biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, hepatic ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) — low anterio resection with hepatic resection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) - Arm A (N=10) | Standard of Care (SOC) - Arm B + Lead in (N=16)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 7 (11)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 7 (13)
Alkaline phosphatase increased (Investigations) | 2 (2) | 7 (11)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (15) | 9 (25)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 6 (8)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 7 (12)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Jaundice (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (4)
Blurred vision (Eye disorders) | 1 (1) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Cardiac disorders - Other, Coronary vasospasm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, Tachycardia , infusion reaction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, irregular heart beat (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8)
Creatinine increased (Investigations) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 7 (10) | 7 (8)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (3) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Eye disorders - Other, Cryotherapy (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, right eye redness (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (13) | 10 (23)
Fever (General disorders) | 1 (1) | 9 (14)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 5 (6) | 6 (13)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other, Swelling/tightening (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Glucosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 5 (8)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (8)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (5) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (7) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 5 (15)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, right subclavian port-a-cath (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 5 (10)
Infusion site extravasation (General disorders) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 3 (6) | 10 (14)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Localized edema (General disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (13) | 9 (25)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 6 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (4)
Nausea (Gastrointestinal disorders) | 7 (13) | 9 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, right conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system disorders - Other, neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 7 (15) | 5 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 10 (16)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (18) | 7 (18)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 10 (12) | 9 (9)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7) | 11 (17)
Platelet count decreased (Investigations) | 5 (10) | 5 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (6) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, cold induced pharyngolaryngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 3 (4)
Skin and subcutaneous tissue disorders - Other, Excoriation and bleeding at the colostomy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Soft tissue infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 4 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Colonoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Kyphoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Sigmoidoscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) — Small bowel resection, enterotomy repair, exploratory laparotomy with lysis of adhesions
Surgical and medical procedures - Other, Stent change (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, stent ERCP (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (5)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (2) | 3 (5)
White blood cell decreased (Investigations) | 7 (10) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03050814/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03050814/ICF_001.pdf